CLINICAL TRIAL: NCT07025733
Title: Clinical Outcomes Related to Treatment of Ankle Injury Using Semiconductor Embedded Therapeutic Socks: A Randomized, Prospective, Double Blinded Clinical Study
Brief Title: Semiconductor Embedded Socks for Ankle Sprains
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado Health (Other); INCREDIWEAR HOLDINGS, INC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-1786
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Ankle Sprain
Keywords: ankle sprain; ligamentous sprain; avulsion fracture; distal fibula fracture
MeSH Terms: conditions — Ankle Injuries; Fractures, Avulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semiconductor Embedded Sock (Experimental)
  Interventions: Device: Semiconductor Embedded Sock
- Control Compression Sock (Placebo Comparator)
  Interventions: Device: Control Compression Sock

INTERVENTIONS:
Device: Semiconductor Embedded Sock — Semiconductor Embedded sock will be given to this intervention arm
  Arms: Semiconductor Embedded Sock
Device: Control Compression Sock — Control sock that is just compression sock
  Arms: Control Compression Sock

SUMMARY:
The goal of this clinical trial is to determine if semiconductor fabric embedded in socks can improve healing after non operative ankle sprains. The main questions it aims to answer are:

1. How does semiconductor embedded sock effect outcomes in patients undergoing rehabilitation from ankle injury?
2. How does semiconductor embedded socks effect injury symptoms and function throughout the course of treatment?

Researchers will compare semiconductor embedded socks with typical compression socks to determine differences in healing.

Participants will be given the socks and be asked to wear them throughout the healing process and record symptoms and functional measures.

DETAILED DESCRIPTION:
STUDY SUMMARY Injuries to the foot and ankle are highly prevalent, with great susceptibility to various injury types due to high usage and complex structural makeup. Ankle injuries are responsible for over 1 million Emergency Room visits each year, and ankle sprains are seen at an incidence of up to 19.0 - 26.6 per 1000 person-years. Approximately 2 million ankle sprains occur annually in the United States alone, and the incidence of re-injury is high, between 12 - 47% of reported ankle sprains are recurrent following initial injury. Ankle sprains are the most commonly presenting sports-related injury each year. Lateral ankle sprains are the most commonly reported type of ankle sprains compared to syndesmotic and medial sprains, and females are at greater risk of sustaining an ankle sprain compared with male counterparts.

Symptoms include pain, swelling, instability and tenderness. Ankle sprains are generally considered treatable and return to activity and sport are typically expected to be successful with proper rehabilitation adherence and measures taken to reduce risk of complication.

The proposed study seeks to evaluate the effectiveness of a non-compressive, therapeutic socks throughout a 12-week course of rehabilitation for non-surgically treated ankle sprain or fracture injury. Outcome measures will be collected at standard intervals up to 1 year to evaluate effectiveness of treatment.

BACKGROUND Treatment approaches for ankle injuries are dictated by the injury type and severity, and include early immobilization, bracing and splinting, return to mobilization as tolerated, rehabilitation strengthening exercises, stabilizing shoes or devices, and pain medication.

Evidence from Lamb, et. al supports a period of up to 14 days of immobilization in a below-knee cast or Aircast instead of a tubular compression bandage and demonstrates improved quality of ankle function after 3 months.

Unlike compression products, the therapeutic socks which will be used in this study are made with semiconductor embedded fabric. The socks increase blood circulation through activation of the embedded elements with heat of the body, and releases mid and far infrared waves as well as negative ions. Both infrared waves and negative ions are biologically active and mediate inflammatory and pain pathways in the body. The technology has also been shown to:

* Increase blood flow and velocity
* Reduce osteoarthritis pain
* Reduce effusion post total knee arthroplasty
* Improve chondrogenic differentiation in vitro
* Improve muscle recovery
* Increase blood speed by up to 22% at rest
* Improve functional outcomes

The benefits of the Infrared Wave and Negative Ion therapy include:

* Inhibition of Cox-2 and Prostaglandins in the lipopolysaccharide (LPS)-moderated pain pathway
* Up-regulation of heat shock protein
* Mediated Nitric oxide production
* Increased activity of voltage-gated ion channels
* Increased activity of mechanosensitive ion channels
* Polarization of cell surface membranes
* Protecting muscle damage
* Scavenging of Reactive Oxygen Species (ROS)
* Improved thermoregulation

The semiconductor embedded fabric emits mid-level and far infrared waves and negative ions. Delivery of infrared waves and negative ions to the tissue increases circulation of both blood and lymph, facilitates the anti-inflammatory nitric oxide (NO) cascade by accelerating the binding of calcium (Ca2+) to calmodulin (CaM). NO provides several healing factors to the body, increasing blood and lymphatic flow6. Additionally, NO down-regulates interleukin-1 beta (IL1β) and inducible nitric oxide synthase (iNOS) in certain cell types, which leads to reduced cyclooxygenase-2 (COX-2) and prostaglandins - molecules responsible for causing inflammation and pain. Unlike other systemic COX-2 inhibitors such as nonsteroidal anti-inflammatory drugs (NSAIDs), targeted infrared and negative ion therapy stimulate localized reaction pathways, thereby reducing pain and inflammation.

This study seeks to identify subjective and objective outcomes for management of ankle sprain, non-operative distal fracture or avulsion fracture injuries through application of semiconductor embedded socks to the affected area.

OBJECTIVES

1. Determine the effect of the semiconductor embedded sock on outcomes in patients undergoing rehabilitation from ankle injury.
2. Evaluate the change in ankle injury symptoms and function in patients throughout the course of treatment with the semiconductor embedded sock.

ELIGIBILITY:
Inclusion Criteria:

* Ankle sprain, avulsion fracture, distal fibular fracture
* Pain for at least 1 day
* Patients 18-69 years old

Exclusion Criteria:

* Patients with neurological conditions
* Patients with prior surgical treatment of lower limb injury
* Patients with chronic pain conditions
* Patient with auto-immune or auto-inflammatory disease
* Patients with tobacco use in last 90 days
* Patients with history of metabolic disorders
* Patients with open wound at area of application
* Patients with acute or systemic infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
FAOS Score | 6 months
  Improved patient function compared to placebo group as determined by pre-treatment and post-treatment Patient Specific Foot Function Index Foot and Ankle Outcome Score (FAOS) compared to placebo group. Range of Scores: [0-100], higher scores indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Alfonso, MD, Principal Investigator — University of Colorado Department of Orthopedics
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No